CLINICAL TRIAL: NCT05604807
Title: From the Classroom to the Rural Community: Engaging Nursing College Students to Create a Dementia-friendly Community Using Virtual Reality and World café Teaching Strategies
Brief Title: Dementia-friendly Community Training Using Virtual Reality Among College Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tzu Chi University (Other)
Responsible Party: Principal Investigator, Huei-Chuan Sung, Associate professor, Tzu Chi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202107ES024
Record Dates: First submitted 2022-10-31; First posted 2022-11-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: two-group randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dementia course with virtual reality (Experimental): Dementia course with virtual reality consists of dementia virtual reality activity, intergenerational learning, world café teaching method and community practice
  Interventions: Other: Dementia course with virtual reality
- Dementia course with no virtual reality (Active Comparator): Dementia course with no virtual reality consists of intergenerational learning, world café teaching method and community practice with no dementia virtual reality activity.
  Interventions: Other: Dementia course with no virtual reality

INTERVENTIONS:
Other: Dementia course with virtual reality — dementia virtual reality activity, intergenerational learning, world café teaching method and community practice
  Arms: Dementia course with virtual reality
Other: Dementia course with no virtual reality — dementia course, intergenerational learning, world café teaching method and community practice
  Arms: Dementia course with no virtual reality

SUMMARY:
This study aims to evaluate the effectiveness of a dementia course using virtual reality, world café teaching method and community practice on knowledge of dementia and dementia-friendly community, attitude toward dementia, and empathy toward people with dementia among nursing college students.

DETAILED DESCRIPTION:
This two-group randomised controlled trial aims to evaluate the effectiveness of a dementia course using virtual reality on knowledge of dementia and dementia-friendly community, attitude toward dementia, and empathy toward people with dementia among nursing college students.

The interventional group will receive the dementia course consists of dementia virtual reality activity, intergenerational learning, world café teaching method and community practice.

The control group will only receive the dementia course with intergenerational learning, world café teaching method and community practice but no dementia virtual reality activity.

Both groups will be assessed for their dementia knowledge, attitudes, empathy and knowledge of dementia-friendly community at baseline, week 8, and week 18.

ELIGIBILITY:
Inclusion Criteria:

* college nursing students with age ranged from 19 to 40 years,
* Taiwanese nationality,
* Sophomore and above
* provide informed consent to participate in the study.

Exclusion Criteria:

college nursing students who do not meet the inclusion criteria

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-17 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Dementia Knowledge Assessment Scale (DKAS) | baseline
  score of knowledge about dementia (0~50) higher scores indicate more knowledge about dementia
Dementia Knowledge Assessment Scale (DKAS) | week 8
  score of knowledge about dementia (0~50) higher scores indicate more knowledge about dementia
Dementia Knowledge Assessment Scale (DKAS) | week 18
  score of knowledge about dementia (0~50) higher scores indicate more knowledge about dementia
Approaches to Dementia Questionnaire (ADQ) | baseline
  score of attitude toward people with dementia (19~95) higher scores indicate more positive attitude towards dementia
Approaches to Dementia Questionnaire (ADQ) | week 8
  score of attitude toward people with dementia (19~95) higher scores indicate more positive attitude towards dementia
Approaches to Dementia Questionnaire (ADQ) | week 18
  score of attitude toward people with dementia (19~95) higher scores indicate more positive attitude towards dementia
Jefferson Scale of Empathy (JSE) | baseline
  score of empathy (20~140) higher scores indicate more empathy for people with dementia
Jefferson Scale of Empathy (JSE) | week 8
  score of empathy (20~140) higher scores indicate more empathy for people with dementia
Jefferson Scale of Empathy (JSE) | week 18
  score of empathy (20~140) higher scores indicate more empathy for people with dementia

SECONDARY OUTCOMES:
Dementia-friendly community questionnaire | baseline
  score of knowledge on dementia-friendly community (0~20) higher scores indicate more knowledge about dementia-friendly community
Dementia-friendly community questionnaire | week 8
  score of knowledge on dementia-friendly community (0~20) higher scores indicate more knowledge about dementia-friendly community
Dementia-friendly community questionnaire | week 18
  score of knowledge on dementia-friendly community (0~20) higher scores indicate more knowledge about dementia-friendly community

CONTACTS AND LOCATIONS:
Locations (1):
- Tzu Chi University, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No